CLINICAL TRIAL: NCT04897139
Title: Phase II Clinical Trial of Flu-Bu-Mel-E (Fludarabine, Busulfan, Melphalan and Etoposide) as Conditioning Regimen for Patients With Lymphoid Malignancies Undergoing Allogeneic Stem Cell Transplantation
Brief Title: Flu-Bu-Mel Based Conditioning Regimen for Patients With Lymphoid Malignancies Undergoing Allo-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, BMT program, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-Lym-2021
Record Dates: First submitted 2021-05-19; First posted 2021-05-21 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Lymphoid Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): treatment arm
  Interventions: Drug: Flu-Bu-Mel-E

INTERVENTIONS:
Drug: Flu-Bu-Mel-E — Fludarabine 150mg/m2, busulfan 6.4mg/kg, melphalan 100mg/m2 and etoposide 600mg/m2

SUMMARY:
In this phase II clinical trial, we evaluate the efficacy and feasibility of conditioning regimen of fludarabine 150mg/m2, busulfan 9.6mg/kg, melphalan 100mg/m2 and etoposide 800mg/m2 in patients with lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* lymphoid malignancies
* donor available: HLA matched sibling, unrelated donor or haplo-identical related donor.
* patients with ECOG <3

Exclusion Criteria:

* inform consent not provided
* ECOG >=3
* poor liver function (enzyme >2N or bilirubin >2N)
* poor renal function (Scr >2N)
* poor cardiac function (EF <45%)

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 1 year after allo-HSCT
  event defined as disease progression, relapse or death of any causes

SECONDARY OUTCOMES:
Overall survival | 1 year after allo-HSCT
  event defined as death of any causes
Non relapse morality | 1 year after allo-HSCT
  event defined as death of any causes except for disease progression or relapse
Relapse | 1 year after allo-HSCT
  event defined as disease progression or relapse
GVHD-free or relapse-free survival | 1 year after allo-HSCT
  event defined as disease progression or relapse, death of any cause, grade III-IV aGVHD or moderate to severe cGVHD

CONTACTS AND LOCATIONS:
Overall Officials: Jiong HU, Principal Investigator — Ruijin Hospital
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, China